CLINICAL TRIAL: NCT03525223
Title: Impact of Changes in Dialysis Sodium Concentration on Tissue Sodium Storage in Hemodialysis Patients
Brief Title: Modulation of Tissue Sodium in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DNa
Record Dates: First submitted 2018-04-24; First posted 2018-05-15 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2020-11

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: 23Na MRI
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dialysate [Na+] 138 mmol/l (Active Comparator): Intervention: Change of dialysate [Na+] from 138 mmol/l to 142 mmol/l The dialysate [Na+] will be increased by 2 mmol/l per week and kept constant for 5 weeks (altogether 6 weeks). Before and after intervention tissue [Na+] will be determined by sodium MRI. Additionally body fluid distribution (by bioimpedance spectroscopy) and central arterial pressure wave form, pulse wave velocity as well as flow-mediated vasodilatation will be assessed.
  Interventions: Procedure: Change of dialysate [Na+]
- dialysate [Na+] 142 mmol/l (Active Comparator): Intervention: Change of dialysate [Na+] from 142 mmol/l to 135 mmol/l The dialysate [Na+] will be decreased by 2 mmol/l per week for 3 weeks and by 1mmol/l for 1 further week. Afterwards the dialysate [Na+] will be kept constant for 5 weeks (altogether 8 weeks). Before and after intervention tissue [Na+] will be determined by sodium MRI. Additionally body fluid distribution (by bioimpedance spectroscopy) and central arterial pressure wave form, pulse wave velocity as well as flow-mediated vasodilatation will be assessed.
  Interventions: Procedure: Change of dialysate [Na+]

INTERVENTIONS:
Procedure: Change of dialysate [Na+] — Stepwise modulation of dialysate sodium concentration by 1-2 mmo/l per week

SUMMARY:
Salt (NaCl) intake is implicated in causing hypertension and cardiovascular disease, the commonest cause of death worldwide. The investigators recently established that Na+ is stored in tissues, bound to glycosaminoglycans (GAGs) in skin and muscle. The resulting local hypertonicity leads to immune cell-driven induction of local tissue electrolyte clearance via modulation of cutaneous lymph capillary density. To visualize these complex processes in man directly, the investigators established Na+ magnetic resonance imaging (23Na-MRI) and investigated Na+ stores in hemodialysis (HD) patients. Hemodialysis patients were sodium-"overloaded" and HD treatment lowered tissue Na+ stores in this study. The observed effects were highly variable and independent of Na+ or water removal from the body during a dialysis session. Tissue Na+ mobilization correlated with circulating vascular endothelial growth factor-C (VEGF-C). The investigators believe that excessive Na+ storage is a reversible condition and therefore susceptible for therapeutic interventions. The investigators hypothesize that lowering dialysate Na+ concentration may favorably affect accelerated tissue Na+ accumulation in hemodialysis patients. Besides, improved tissue Na+ storage, osmostress-induced as well as pro-inflammatory immune cell response should be affected by such a revised dialysis management.

DETAILED DESCRIPTION:
To evaluate effects of moderate reduction of dialysate Na+ concentration on tissue Na+ content the investigators intend to recruit 40 hemodialysis patients, who will be offered a therapeutic change of their dialysate Na+ concentration. After detection of tissue Na+ content using 23Na-MRI technique, the applied dialysate [Na+] will be initially increased stepwise by 2 mmol/l per week from 138 to 142 mmol/l and maintained for a period of 5 weeks. After another 23Na-MRI measurement, dialysate [Na+] will then be lowered stepwise by 1-2 mmol/l per week to a minimum of 135 mmol/l, which will be also maintained for a period of 5 weeks followed by a final 23Na-MRI assessment.

Hypothesis: Reduction of dialysate Na+ concentration will decrease tissue sodium storage.

Additionally, the investigators will assess changes in body fluid distribution by bioimpedance spectroscopy. Furthermore, vascular compliance in response to the modulation of dialysate [Na+] and its correlation with tissue Na+ will be assessed. To investigate the immune response to tissue Na+ accumulation, the osmostress-induced as well as pro-inflammatory immune cell response of isolated monocytes will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Stage 5D, hemodialysis performed for at least 6 months, three times hemodialysis per week, signed informed consent

Exclusion Criteria:

* Pregnancy, severe heart failure (NYHA III - IV), severe liver disease (CHILD C), acute infection, pacemaker or other non-MRI suitable conditions, hyponatremia < 132 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Tissue sodium content | 14 weeks
  Tissue sodium content measured by 23Na MRI

SECONDARY OUTCOMES:
Lymphangiogenic profile | 14 weeks
  Serum VEGF-C and sFLT4 levels will be determined
Body fluid distribution (extracellular and intracellular water) | 14 weeks
  Change in body fluid distribution will be assessed by body composition monitor (bioimpedance spectroscopy)
Pulse wave analysis and pulse wave velocity | 14 weeks
  Change in central arterial pressure wave form and pulse wave velocity will be analyzed by SphygmoCor
Flow-mediated vasodilatation (FMD) | 14 weeks
  Measurement of vasodilatation and thereby arterial stiffness by a semi-automated ultrasound System (UNEXEF)
Immune response to tissue Na+ accumulation | 14 weeks
  Blood monocytes will be isolated and their osmotic and inflammatory response will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kopp, MD, Principal Investigator — Nephrology Department, University Erlangen, Germany
Locations (1):
- Nephrology Department, University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlmann A, Dorfelt K, Eicher F, Linz P, Kopp C, Mossinger I, Horn S, Buschges-Seraphin B, Wabel P, Hammon M, Cavallaro A, Eckardt KU, Kotanko P, Levin NW, Johannes B, Uder M, Luft FC, Muller DN, Titze JM. Magnetic resonance-determined sodium removal from tissue stores in hemodialysis patients. Kidney Int. 2015 Feb;87(2):434-41. doi: 10.1038/ki.2014.269. Epub 2014 Aug 6. PMID 25100048
- [Background] Kopp C, Linz P, Maier C, Wabel P, Hammon M, Nagel AM, Rosenhauer D, Horn S, Uder M, Luft FC, Titze J, Dahlmann A. Elevated tissue sodium deposition in patients with type 2 diabetes on hemodialysis detected by 23Na magnetic resonance imaging. Kidney Int. 2018 May;93(5):1191-1197. doi: 10.1016/j.kint.2017.11.021. Epub 2018 Feb 15. PMID 29455909
- [Background] Titze J, Dahlmann A, Lerchl K, Kopp C, Rakova N, Schroder A, Luft FC. Spooky sodium balance. Kidney Int. 2014 Apr;85(4):759-67. doi: 10.1038/ki.2013.367. Epub 2013 Oct 9. PMID 24107854